CLINICAL TRIAL: NCT00523809
Title: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation With Bevacizumab for Advanced Solid Tumor
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation With Bevacizumab for Advanced Solid Tumor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0873
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Breast Cancer; Ovarian Cancer; Stem Cell Transplantation; Bevacizumab; Fludarabine; Melphalan; Avastin; Thymoglobulin; ATG; Antithymocyte Globulin; Allogeneic Hematopoietic Stem Cell Transplantation; AHSCT
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; fludarabine; fludarabine phosphate; Melphalan; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + Fludarabine + Melphalan (Experimental): Bevacizumab 10 mg/kg intravenous (IV) on Day 1; Fludarabine 25 mg/m^2 IV Daily over 5 Days; Melphalan 70 mg/m^2 IV Daily over 2 Days; Thymoglobulin 0.5 mg/kg IV on Day - 3, 1.5 mg/kg IV on Day - 2, and 2 mg/kg IV on Day -1; plus Allogeneic Hematopoietic Stem Cell Transplantation on Day 8.
  Interventions: Drug: Bevacizumab; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Fludarabine; Drug: Melphalan; Drug: Thymoglobulin

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg IV Daily Over 30 Minutes for 1 Day
  Other Names: Avastin™; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Stem Cell Transplantation on Day 8.
  Other Names: NST
Drug: Fludarabine — 25 mg/m^2 IV Daily Over 30 Minutes for 5 Days
  Other Names: Fludarabine Phosphate
Drug: Melphalan — 70 mg/m^2 IV Daily Over 30 Minutes for 2 Days
Drug: Thymoglobulin — 0.5 mg/kg IV on Day - 3, 1.5 mg/kg IV on Day - 2, and 2 mg/kg IV on Day -1.
  Other Names: ATG; Antithymocyte Globulin

SUMMARY:
The goal of this clinical research study is to learn if giving Avastin (bevacizumab) with standard chemotherapy and a blood stem cell transplant, in patients with an advanced solid tumor, can help to shrink the tumor or slow its growth. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

The combination of standard chemotherapy drugs (fludarabine and melphalan) used for this study may help to improve the chances of your body accepting the stem cell transplant. Fludarabine is designed to make cancer cells less able to repair damaged DNA (the genetic material of cells) and weaken the immune system so that stem cells can stay in your body. Melphalan is designed to damage the cancer cells' DNA.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will have a central venous catheter inserted. A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

You will receive chemotherapy with bevacizumab, fludarabine, and melphalan in order to prepare for the stem cell transplant.

On Day 1, you will receive bevacizumab through a needle in your vein over 30 minutes.

On Days 2-6, you will receive fludarabine by vein over 30 minutes.

On Day 5-6, you will receive melphalan by vein over 30 minutes.

On Day 7, you will receive no study drugs.

Stem Cell Transplant and Post-Transplant Drug Administration:

On Day 8, you will have a stem cell transplant. Your study doctor will explain this procedure to you in more detail and you will sign a separate consent form.

After the transplant, you will receive the drugs tacrolimus and methotrexate. Tacrolimus and methotrexate are used to prevent graft versus host disease (GVHD), a condition that occurs when the transplanted cells attack the normal cells in the body.

Tacrolimus will be given by vein non-stop (24 hours a day) until you are able to take medications by mouth. Once you are able to take medications by mouth, your doctor will tell you how and when to take the oral medication. You will receive tacrolimus for 2-3 months. During the last month that tacrolimus is given, the dose will be lowered gradually.

Methotrexate will be given by vein over a few seconds on Days 9, 11, and 14. An additional dose of methotrexate will be given on Day 19 if your donor is your parent, child, or an unrelated family member.

If GVHD does occur, the GVHD will be treated with methylprednisolone by vein or by mouth, as needed. You may also be given steroid cream to use on the skin, if needed.

Starting at least 3 weeks after the transplant, as soon as your blood counts recover, you will receive bevacizumab every 2 weeks by vein over 30 minutes.

Post-Transplant Procedures:

You must stay in the hospital for about 3-4 weeks beginning on Day 1. While you are in the hospital, blood (about 2 teaspoons) will be drawn for routine tests every day.

You must stay in the Houston area for about 100 days after the transplant. Once a month during the 100 days after the transplant, and then every 3 months for the first year, you will have scans to check the status of the disease. The study doctor will decide which scans are necessary (chest x-rays, CT scans, and/or bone scans). You may also have a bone marrow aspirate and biopsy at these times. The bone marrow aspirate and biopsy would only be performed if your bone marrow was shown to be involved with the disease at the time of screening.

If the disease is still present at 2 months after the transplant, and you do not have GVHD, you will stop receiving tacrolimus within 2 weeks. After that, if the disease is still present after another 6 weeks, and you do not have GVHD, you may receive an infusion of donor lymphocytes (a type of white blood cell) by vein over about 30 minutes. This treatment with white blood cells may be repeated 2 more times with 6 weeks between each infusion.

Length of Study:

You will be taken off-study after 1 year.

Follow-Up Visits:

You will have follow-up visits as per standard of care.

This is an investigational study. The use of bevacizumab in transplant patients is not FDA approved. Melphalan and fludarabine are FDA approved and commercially available for transplant patients. Up to 18 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. From Age 18 to Age </= 65 years old.
2. Patients must have one of the following diseases. 1) metastatic breast cancer which achieved a tumor response (complete response (CR) or partial response (PR)) by pre-transplant therapy. For bone only metastatic breast cancer, a tumor response of stable disease (SD) is accepted. 2) low grade advanced ovarian cancer 3) high grade advanced ovarian cancer which achieved antitumor response (CR or PR) by pre-transplant therapy.
3. Zubrod performance status </= 1.
4. An HLA-matched (6/6 matches) related donor or unrelated donor (8/8 matches) willing and able to donate peripheral blood stem cell (PBSC) or bone marrow and/or lymphocytes by conventional techniques.
5. Requirement of prior treatment. For metastatic renal cell carcinoma (RCC) two prior treatments, which include targeted therapy (e.g. Sorafenib and Stutent). For breast and ovarian cancer, one prior treatment which include chemotherapy.
6. Adequate major organ functions.
7. Signed informed consent.
8. Left ventricular ejection fraction >/= 45%. Cardiology clearance is needed if the patient has left ventricular ejection fraction of < 45%, uncontrolled arrhythmias, or symptomatic cardiac disease.
9. Forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC), and carbon monoxide diffusing capacity (DLCO) >/= 50% of predicted value. Pulmonary clearance is needed if the patient has FEV1, FVC, or DLCO < 50% of predicted valued or any symptomatic pulmonary disease.
10. Serum creatinine </= 2.0 mg/dL, or creatinine clearance > 40 mL/min.
11. Serum bilirubin </= 1.5 mg/dL, and serum glutamic-pyruvic transaminase (SGPT) </= 3 * upper limit of normal.

Exclusion Criteria:

1. Prior history of allogeneic stem cell transplantation.
2. Life expectancy is severely limited by concomitant illness.
3. Clinically significant active infections.
4. HIV infection.
5. Chronic active hepatitis.
6. Pregnant or lactating women.
7. Presence of, or prior history of multiple brain metastasis. If patient has prior single brain metastasis treated with complete surgical resection or stereotactic radiation therapy, radiological imaging has to demonstrate no recurrence or no brain edema for at least 6 months from the end of the treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 30. 2007 through November 2, 2010. All recruitment was done at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Bevacizumab + Fludarabine + Melphalan
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + Fludarabine + Melphalan
Number analyzed (Participants) | 5
Age Continuous [Median (Full Range); unit: years] | 55 [45 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Number or participants with no disease progression or death for any reason during first 100 days following transplantation. Participants followed every 3 months for first year.
Time Frame: 100 days after transplant
Population: Study objectives were not meet, analysis was not performed.
Arm/Group | Bevacizumab + Fludarabine + Melphalan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year and 7 months
Arm/Group | Bevacizumab + Fludarabine + Melphalan
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Fludarabine + Melphalan (N=5)
Diverticulitis (Gastrointestinal disorders) | 1
Death (Investigations) | 1
Cardiac toxicity, reduced ejection fraction (Cardiac disorders) | 1
Headache (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Fludarabine + Melphalan (N=5)
Vaginal bleed (Reproductive system and breast disorders) | 1
Hot flash (Reproductive system and breast disorders) | 1
Vaginal itch (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Mild breast pain (Reproductive system and breast disorders) | 1
Face swelling (Reproductive system and breast disorders) | 1
Mild depression (Psychiatric disorders) | 1
Headache (General disorders) | 1
Abdominal tenderness (Investigations) | 1
Insomnia (Psychiatric disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No